CLINICAL TRIAL: NCT06449144
Title: The Effect of Mindfulness Training on Postoperative Pain - A Solomon Four Group Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Principal Investigator, Hülya Saray Kılıç, Assisstant Professor, Bilecik Seyh Edebali Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BilecikSeyhEU1
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Pain; Inguinal Hernia Repair; Mindfulness Training
Keywords: inguinal hernia repair; postoperative pain; mindfulness training; intrusion of pain; fear of pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients who are decided to undergo surgery and meet the inclusion criteria will be informed about the study and invited to participate. Patients who agree to participate in the study will be randomly divided into groups. Block randomization will be applied because the participants will receive preoperative and postoperative care in the same clinic and are likely to interact with each other. Awareness training will be given face-to-face by the investigators 24 hours before surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- mindfulness education with pre-test group (Experimental): 24 hours before surgery, patients will be administered the sociodemographic information form, the fear of pain scale and the cognitive intrusion of pain scale. Subsequently, awareness training will be given to the patients. 24 hours after surgery, surgical information form, fear of pain scale and cognitive intrusion of pain scale will be administered.
  Interventions: Other: Mindfulness education
- mindfulness education without pre-test group (Experimental): 24 hours before surgery awareness training will be given to the patients. 24 hours after surgery, surgical information form, fear of pain scale and cognitive intrusion of pain scale will be administered.
  Interventions: Other: Mindfulness education
- control with pre-test group (No Intervention): 24 hours before surgery, patients will be administered the sociodemographic information form, the fear of pain scale and the cognitive intrusion of pain scale. 24 hours after surgery, surgical information form, fear of pain scale and cognitive intrusion of pain scale will be administered.
- control without pre-test group (No Intervention): 24 hours after surgery, surgical information form, fear of pain scale and cognitive intrusion of pain scale will be administered.

INTERVENTIONS:
Other: Mindfulness education — The mindfulness-based stress reduction method was examined and a two-step mindfulness education is planned. To reveal the experience of pain: It was planned to conduct interviews with the participants to realize what they think about the pain they have experienced before or what they think about the pain they have experienced here and now, what emotions they have, and their experiences related to their coping processes with pain. Participants will be encouraged to notice negative thoughts that could impact their coping with pain negatively, and they will be provided with education on the benefits of managing the process of changing these negative thoughts. Attempts will be made to establish positive thinking. Attention: Recognizing the relationship between pain sensation and attention and encouraging its expression is included in the intervention. Information on distraction was given and two exercises we planned to increase the level of awareness.
  Arms: mindfulness education with pre-test group; mindfulness education without pre-test group

SUMMARY:
The goal of this clinical trial is to learn if mindfulness education works to reduce pain after inguinal hernia operation in adults. The main questions it aims to answer are:

Does mindfulness education reduce the pain level after inguinal hernia operation? Does mindfulness education reduce the pain intrusion level after inguinal hernia operation? Does mindfulness education reduce the fear of pain level after inguinal hernia operation?

Participants will:

Pain level, pain intrusion and fear of pain levels will be determined 24 hours before surgery.

Awareness training will be given before surgery. Pain level, pain intrusion and fear of pain levels will be determined 24 hours after surgery.

DETAILED DESCRIPTION:
Cognitive behavioral therapy and mindfulness-based therapies are successful practices in reducing anxiety and psychological distress (Ghielen et al. 2019). Mindfulness training includes teaching a range of meditation techniques as well as how to focus on the present moment in daily activities (Monshat, K., & Castle, D. J., 2012). Mindfulness training given to patients undergoing hip replacement surgery has been shown to reduce postoperative pain and improve their physical functioning (Dowsey et al., 2019). Similarly, it has been reported that mindfulness training given to patients who will undergo knee and hip replacement before surgery can prevent postoperative pain and opioid use (Hanley et al., 2021). In a study, mindfulness training used in the management of pain after lumbar disc herniation surgery was found to be useful in managing postoperative pain (Juneyoung et al., 2019). Aromatherapy with lavender oil was found to be effective in reducing pain after inguinal hernia surgery (Bagheri et al., 2020). This suggests that in addition to pharmacological pain management, non-pharmacological methods are also effective in pain management and can be used. In a meta-analysis evaluating the effectiveness of mindfulness-based interventions in acute pain, it was found that there was a lack of good quality evidence for the effectiveness of mindfulness-based interventions in reducing pain severity in clinical or experimental settings (Shires et al., 2020). It is stated that more rigorous large-scale studies conducted with pain populations are needed before cognitive behavioral therapies can be definitively recommended as first-line treatment for acute or chronic pain (McClintock et al., 2021). Therefore, our study was planned to determine the effect of preoperative awareness training on postoperative pain in patients undergoing inguinal hernia repair surgery.

ELIGIBILITY:
Inclusion Criteria:

* agreeing to participate in research
* planned inguinal hernia surgery with mash
* to be able to read and understand Turkish
* ASA I-III

Exclusion Criteria:

* bilateral or revision inguinal hernia surgery planned
* having a mental illness
* use of opioid-derived medication in the last month
* wanting to leave at any stage of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Pain level | 24 hours after surgery
  The Visual Analogue Scale (VAS) of the patients who took the mindfulness education is decreased compared to those who do not. A score between 0 and 10 is taken from the VAS. It is good that the score from the VAS has decreased.

SECONDARY OUTCOMES:
Fear of Pain | 24 hours after surgery
  Fear of pain of the patients who took the mindfulness education is decreased compared to those who do not. A score between 1 and 5 is taken from the scale. It is good that the score from the scale score has decreased.
Intrusion of pain | 24 hours after surgery
  Intrusion of pain of the patients who took the mindfulness education is decreased compared to those who do not. A score between 0 and 6 is taken from the scale. It is good that the score from the scale has decreased.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Bilecik Eğitim ve Araştırma Hastanesi, Bilecik
  - Bilecik Şeyh Edebali University, Bilecik

IPD SHARING:
Plan to Share IPD: Undecided
A decision will be made after consultation with other researchers.

REFERENCES:
- [Background] Yi JL, Porucznik CA, Gren LH, Guan J, Joyce E, Brodke DS, Dailey AT, Mahan MA, Hood RS, Lawrence BD, Spiker WR, Spina NT, Bisson EF. The Impact of Preoperative Mindfulness-Based Stress Reduction on Postoperative Patient-Reported Pain, Disability, Quality of Life, and Prescription Opioid Use in Lumbar Spine Degenerative Disease: A Pilot Study. World Neurosurg. 2019 Jan;121:e786-e791. doi: 10.1016/j.wneu.2018.09.223. Epub 2018 Oct 9. PMID 30312812
- [Background] Yang J, Lo WLA, Zheng F, Cheng X, Yu Q, Wang C. Evaluation of Cognitive Behavioral Therapy on Improving Pain, Fear Avoidance, and Self-Efficacy in Patients with Chronic Low Back Pain: A Systematic Review and Meta-Analysis. Pain Res Manag. 2022 Mar 19;2022:4276175. doi: 10.1155/2022/4276175. eCollection 2022. PMID 35345623
- [Background] Hanley AW, Garland EL, Zingg RW. Mindfulness-based waiting room intervention for osteopathic manipulation patients: a pilot randomized controlled trial. J Osteopath Med. 2021 Feb 24;121(4):337-348. doi: 10.1515/jom-2020-0186. PMID 33694345
- [Background] Dowsey M, Castle D, Knowles S, Monshat K, Salzberg M, Nelson E, Dunin A, Dunin J, Spelman T, Choong P. The effect of mindfulness training prior to total joint arthroplasty on post-operative pain and physical function: A randomised controlled trial. Complement Ther Med. 2019 Oct;46:195-201. doi: 10.1016/j.ctim.2019.08.010. Epub 2019 Aug 12. PMID 31519279
- [Background] Monshat K, Castle DJ. Mindfulness training: an adjunctive role in the management of chronic illness? Med J Aust. 2012 May 21;196(9):569-71. doi: 10.5694/mja11.10974. PMID 22621147
- [Background] McClintock AS, McCarrick SM, Garland EL, Zeidan F, Zgierska AE. Brief Mindfulness-Based Interventions for Acute and Chronic Pain: A Systematic Review. J Altern Complement Med. 2019 Mar;25(3):265-278. doi: 10.1089/acm.2018.0351. Epub 2018 Dec 5. PMID 30523705
- [Background] Shires A, Sharpe L, Davies JN, Newton-John TRO. The efficacy of mindfulness-based interventions in acute pain: a systematic review and meta-analysis. Pain. 2020 Aug;161(8):1698-1707. doi: 10.1097/j.pain.0000000000001877. PMID 32701830
- [Background] Bagheri H, Salmani T, Nourian J, Mirrezaie SM, Abbasi A, Mardani A, Vlaisavljevic Z. The Effects of Inhalation Aromatherapy Using Lavender Essential Oil on Postoperative Pain of Inguinal Hernia: A Randomized Controlled Trial. J Perianesth Nurs. 2020 Dec;35(6):642-648. doi: 10.1016/j.jopan.2020.03.003. Epub 2020 Jul 21. PMID 32709507
- [Background] Ghielen I, Rutten S, Boeschoten RE, Houniet-de Gier M, van Wegen EEH, van den Heuvel OA, Cuijpers P. The effects of cognitive behavioral and mindfulness-based therapies on psychological distress in patients with multiple sclerosis, Parkinson's disease and Huntington's disease: Two meta-analyses. J Psychosom Res. 2019 Jul;122:43-51. doi: 10.1016/j.jpsychores.2019.05.001. Epub 2019 May 13. PMID 31126411